CLINICAL TRIAL: NCT04706442
Title: Evaluate the Effectiveness and Cost-effectiveness of 'Supportive Parenting App' a Mobile Based Application on Parental and Newborn Outcomes: A Multi-center Randomized Controlled Trial
Brief Title: Effectiveness of 'Supportive Parenting App' on Parental and Newborn Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Shefaly Shorey, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHG DSRB 2019/00875
Record Dates: First submitted 2021-01-07; First posted 2021-01-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Postnatal Depression; Self Efficacy; Parent-Child Relations; Development, Child; Anxiety; Parenting Satisfaction
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard hospital care with follow up + Supportive Parenting App (Experimental): Receive standard hospital care and follow up, and access to the Supportive Parenting App from pregnancy to 6 months postpartum
  Interventions: Other: Supportive Parenting Application
- Standard hospital care with follow up (No Intervention): Receive standard hospital care with follow up

INTERVENTIONS:
Other: Supportive Parenting Application — The Supportive Parenting Application is a theory-based perinatal educational intervention for couples administered through a mobile application. The mobile app consist of knowledge-based content, informational videos and audio, discussion forum, chat groups with peer volunteers, and an experts advice section
  Arms: Standard hospital care with follow up + Supportive Parenting App

SUMMARY:
The Supportive Parenting App is a theory-based perinatal educational intervention for couples administered through a mobile application. The intervention comprise of knowledge-based content, informational videos and audio, discussion forum, peer volunteer chat group, and a frequently asked questions (FAQ) expert advice section.

The aims of the study are to:

1. develop theory-based supportive parenting App (SPA) intervention for both first-time and experienced parents across perinatal period
2. examine its effectiveness on parental outcomes: including maternal depression at 12 months postpartum (primary outcome), paternal depression, parental anxiety, parenting self-efficacy, help - seeking behavior (social support), parental bonding and parenting satisfaction (secondary outcomes); and new-born outcomes: physical, social and emotional developments (secondary outcomes)
3. evaluate SPA's cost-effectiveness as compared to standard perinatal care across major restructured hospitals, and
4. examine the perceptions of parents in receiving this intervention.

When compared with those in the control group receiving standard care:

1. parents receiving SPA intervention will have better- emotional well-being (reduced depression and anxiety);parenting self-efficacy; social support; bonding and satisfaction.
2. new-borns of parents receiving SPA will have better physical, social and emotional development
3. It will be more cost-effective to provide SPA than the standard care

ELIGIBILITY:
Inclusion Criteria:

* able to read and speak English
* have low-risk singleton pregnancy with more than 24 weeks of gestation (age of viability)
* have smartphone with internet access

Exclusion Criteria:

* have physical or mental disorders which would interfere with their ability to participate in the study
* have high-risk pregnancy including placenta-previa major, pre-eclampsia, pregnancy induced hypertension etc.
* have complicated assisted delivery such as vacuum or forceps with 4th degree perineal tear of the mother; and /or
* give birth to a newborn at still-birth or a newborn with congenital anomalies and/or medical complications including pathological jaundice, that required special care in hospital.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Maternal postpartum depression | 1 month postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Maternal postpartum depression | 2 month postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Maternal postpartum depression | 4 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Maternal postpartum depression | 6 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Maternal postpartum depression | 9 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Maternal postpartum depression | 12 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome

SECONDARY OUTCOMES:
Infant physical, social, and emotional development | 6 months postpartum
  Bayley-IV scale Minimum raw score of 0 and maximum score of 258 for 129 items. Higher score indicate better outcome
Infant physical, social, and emotional development | 12 months postpartum
  Bayley-IV scale Minimum score of 0 and maximum score of 258 for 129 items. Higher score indicate better outcome
Infant physical, social, and emotional development | 2 months postpartum
  Ages and Stages Questionnaire - 3 (ASQ-3) 21 items; minimum score of 0 and maximum score of 210, with higher score indicating better outcomes
Infant physical, social, and emotional development | 4 months postpartum
  Ages and Stages Questionnaire - 3 (ASQ-3) 21 items; minimum score of 0 and maximum score of 210, with higher score indicating better outcomes
Infant physical, social, and emotional development | 6 months postpartum
  Ages and Stages Questionnaire - 3 (ASQ-3) 21 items; minimum score of 0 and maximum score of 210, with higher score indicating better outcomes
Infant physical, social, and emotional development | 9 months postpartum
  Ages and Stages Questionnaire - 3 (ASQ-3) 21 items; minimum score of 0 and maximum score of 210, with higher score indicating better outcomes
Infant physical, social, and emotional development | 12 months postpartum
  Ages and Stages Questionnaire - 3 (ASQ-3) 21 items; minimum score of 0 and maximum score of 210, with higher score indicating better outcomes
Paternal depression | 1 month postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Paternal depression | 2 month postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Paternal depression | 4 month postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Paternal depression | 6 month postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Paternal depression | 9 month postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Paternal depression | 12 month postpartum
  Edinburgh Postnatal Depression Scale (EPDS) Minimum score is 0, maximum score is 30, with higher score indicating worse outcome
Parental Anxiety | 1 month postpartum
  State-Trait Anxiety Scale (STAI) minimum score of 20 and maximum score of 80, with higher scores indicating worse outcomes.
Parental Anxiety | 2 month postpartum
  State-Trait Anxiety Scale (STAI) minimum score of 20 and maximum score of 80, with higher scores indicating worse outcomes.
Parental Anxiety | 4 month postpartum
  State-Trait Anxiety Scale (STAI) minimum score of 20 and maximum score of 80, with higher scores indicating worse outcomes.
Parental Anxiety | 6 month postpartum
  State-Trait Anxiety Scale (STAI) minimum score of 20 and maximum score of 80, with higher scores indicating worse outcomes.
Parental Anxiety | 9 month postpartum
  State-Trait Anxiety Scale (STAI) minimum score of 20 and maximum score of 80, with higher scores indicating worse outcomes.
Parental Anxiety | 12 month postpartum
  State-Trait Anxiety Scale (STAI) minimum score of 20 and maximum score of 80, with higher scores indicating worse outcomes.
Parenting self-efficacy | 1 month postpartum
  Parenting Efficacy Scale (PES) Scores range from 10 to 40 with higher scores indicating higher parenting efficacy
Parenting self-efficacy | 2 month postpartum
  Parenting Efficacy Scale (PES) Scores range from 10 to 40 with higher scores indicating higher parenting efficacy
Parenting self-efficacy | 4 month postpartum
  Parenting Efficacy Scale (PES) Scores range from 10 to 40 with higher scores indicating higher parenting efficacy
Parenting self-efficacy | 6 month postpartum
  Parenting Efficacy Scale (PES) Scores range from 10 to 40 with higher scores indicating higher parenting efficacy
Parenting self-efficacy | 9 month postpartum
  Parenting Efficacy Scale (PES) Scores range from 10 to 40 with higher scores indicating higher parenting efficacy
Parenting self-efficacy | 12 month postpartum
  Parenting Efficacy Scale (PES) Scores range from 10 to 40 with higher scores indicating higher parenting efficacy
Perceived social support | 1 month postpartum
  Perceived Social Support for Parenting (PSSP) scale minimum score of 10 and maximum score of 40. Higher score indicate higher perceived support.
Perceived social support | 2 month postpartum
  Perceived Social Support for Parenting (PSSP) scale minimum score of 10 and maximum score of 40. Higher score indicate higher perceived support.
Perceived social support | 4 month postpartum
  Perceived Social Support for Parenting (PSSP) scale minimum score of 10 and maximum score of 40. Higher score indicate higher perceived support.
Perceived social support | 6 month postpartum
  Perceived Social Support for Parenting (PSSP) scale minimum score of 10 and maximum score of 40. Higher score indicate higher perceived support.
Perceived social support | 9 month postpartum
  Perceived Social Support for Parenting (PSSP) scale minimum score of 10 and maximum score of 40. Higher score indicate higher perceived support.
Perceived social support | 12 month postpartum
  Perceived Social Support for Parenting (PSSP) scale minimum score of 10 and maximum score of 40. Higher score indicate higher perceived support.
Parent-Infant bonding | 1 month postpartum
  Parent-to-Infant Bonding Scale scores range from 0 to 24, with higher scores indicating worse bonding
Parent-Infant bonding | 2 month postpartum
  Parent-to-Infant Bonding Scale scores range from 0 to 24, with higher scores indicating worse bonding
Parent-Infant bonding | 4 month postpartum
  Parent-to-Infant Bonding Scale scores range from 0 to 24, with higher scores indicating worse bonding
Parent-Infant bonding | 6 month postpartum
  Parent-to-Infant Bonding Scale scores range from 0 to 24, with higher scores indicating worse bonding
Parent-Infant bonding | 9 month postpartum
  Parent-to-Infant Bonding Scale scores range from 0 to 24, with higher scores indicating worse bonding
Parent-Infant bonding | 12 month postpartum
  Parent-to-Infant Bonding Scale scores range from 0 to 24, with higher scores indicating worse bonding
Parenting satisfaction | 1 month postpartum
  What Being the Parent of a New Baby is Like Questionnaire (WPBL) 11-items, scores range from 0 to 99 with higher scores indicating better parenting satisfaction.
Parenting satisfaction | 2 month postpartum
  What Being the Parent of a New Baby is Like Questionnaire (WPBL) 11-items, scores range from 0 to 99 with higher scores indicating better parenting satisfaction.
Parenting satisfaction | 4 month postpartum
  What Being the Parent of a New Baby is Like Questionnaire (WPBL) 11-items, scores range from 0 to 99 with higher scores indicating better parenting satisfaction.
Parenting satisfaction | 6 month postpartum
  What Being the Parent of a New Baby is Like Questionnaire (WPBL) 11-items, scores range from 0 to 99 with higher scores indicating better parenting satisfaction.
Parenting satisfaction | 9 month postpartum
  What Being the Parent of a New Baby is Like Questionnaire (WPBL) 11-items, scores range from 0 to 99 with higher scores indicating better parenting satisfaction.
Parenting satisfaction | 12 month postpartum
  What Being the Parent of a New Baby is Like Questionnaire (WPBL) 11-items, scores range from 0 to 99 with higher scores indicating better parenting satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Shefaly Shorey, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Alice Lee Centre for Nursing Studies, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shorey S, Thilagamangai, Mathews J, Lim SH, Shi L, Chua JS, Du R, Chan YH, Tan TC, Chee C, Chong YS. Effects of Parental Predictors on Postpartum Depression. West J Nurs Res. 2024 Jul;46(7):517-524. doi: 10.1177/01939459241254774. Epub 2024 Jun 1. PMID 38822693
- [Derived] Shorey S, Chong YS, Shi L, Chua JS; Thilagamangai; Mathews J, Lim SH, Du R, Chan YH, Tan TC, Chee C, Law E. Evaluating the Effects of the Supportive Parenting App on Infant Developmental Outcomes: Longitudinal Study. JMIR Mhealth Uhealth. 2023 Feb 22;11:e43885. doi: 10.2196/43885. PMID 36811952
- [Derived] Shorey S, Law E; Thilagamangai; Mathews J, Lim SH, Shi L, Chua JS, Du R, Chan YH, Tan TC, Chee C, Chong YS. Evaluating the Effectiveness of the Supportive Parenting App on Parental Outcomes: Randomized Controlled Trial. J Med Internet Res. 2023 Jan 16;25:e41859. doi: 10.2196/41859. PMID 36645699